CLINICAL TRIAL: NCT06785805
Title: Relationship Between Disease Severity, Pain, Lower Extremity Strength, Respiratory Functions, Aerobic Capacity and Quality of Life in Individuals With Chronic Venous Insufficiency
Brief Title: Respiratory Functions, Aerobic Capacity and Quality of Life in Chronic Venous Insufficiency
Status: Completed | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Özlem Çınar Özdemir, Prof.Dr, Izmir Democracy University
Other Study IDs: IzmirDemocracy University
Record Dates: First submitted 2025-01-15; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Chronic Venous Insufficiency, CVI
Keywords: disease severity; chronic venous insufficiency; respiratory functions
MeSH Terms: conditions — Blindness, Cortical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with Chronic venous insufficiency: Our prospective randomized controlled planned study named 'Inspiratory Muscle Training in Individuals with Chronic Venous Insufficiency: Randomized Controlled Study', which was approved by Izmir Democracy University Non-Interventional Clinical Research Ethics Committee on 21/06/2023 with the decision number 2023/08-02, was conducted. Although 38 individuals diagnosed with CVI were included in the study, the study was completed with 30 individuals diagnosed with CVI who could complete the 6-week follow-up. In the current study, which is a continuation of the previsious research; It is aimed to analyze the initial measurement results of 38 individuals diagnosed with CVI who were initially included in the study and to contribute these data to the literature with a retrospective cross-sectional study design. Our new hypothesis is based on the examination of the correlation between these initial outcome measurements obtained from our previous study.

SUMMARY:
This study aims to retrospectively examine the dataset obtained from a previously conducted study titled 'Inspiratory muscle training in individuals with chronic venous insufficiency: randomized controlled trial'. The previously conducted study was a study investigating the effectiveness of the application, and the current study aims to clarify the gap in the literature with the relationship between the data obtained from the patients at the beginning of that study. This study will be conducted by re-examining the initial data of another study from which data was collected before and conducting new analyses.

H0: There is no relationship between disease severity, edema, pain, respiratory muscle strength, respiratory functions, aerobic capacity, lower extremity strength or quality of life in individuals with chronic venous insufficiency.

H1: There is a relationship between disease severity, edema, pain, respiratory muscle strength, respiratory functions, aerobic capacity, lower extremity strength or quality of life in individuals with chronic venous insufficiency.

DETAILED DESCRIPTION:
Chronic Venous Insufficiency (CVI) is a term used to describe a disorder that affects the venous system of the lower extremities and results in venous hypertension. Venous pathology develops when venous pressure increases and the return of blood is impaired by various mechanisms. These pathologies are caused by valve insufficiency, venous obstruction or inadequate functioning of the muscle pump. The veins in the calf and the tissues surrounding them form the muscle pump. The muscle pump is responsible for venous blood circulation and is activated by ankle movements. In venous insufficiency, one-way valves and vein walls relax, resulting in muscle pump dysfunction. CVI can cause various pathologies and subjective symptoms such as leg pain and cramps, a feeling of heaviness, edema and skin changes. All these symptoms negatively affect the quality of life depending on the intensity of pain, severity of edema and the presence of inflammation. In CVI, the limitation of ankle movement is one of the factors that increase edema and venous severity. Fibrotic tissue formations in the lower extremity cause limitation in ankle movements. It should not be forgotten that functionality and quality of life are closely related phenomena, as the physical activity levels and functional capacity deterioration of people with chronic venous insufficiency increase, the quality of life decreases, which further worsens the prognosis of the disease. Complications of CVI impair the person's ability to participate in social or routine occupational activities, reduce working capacity, and ultimately increase the economic burden on the person and the family. Chronic venous diseases are a common condition that causes great socioeconomic effects due to their high prevalence. 32% of women and 40% of men have varicose veins. In addition, any type of venous disease affects 40-50% of men and 50-55% of women. CVI risk factors include heredity, pregnancy, aging, thrombosis, connective tissue laxity, inactivity, excessive weight, use of high-heeled shoes, standing for long periods, wearing tight clothes, being a woman, geographical effects and improper eating habits. Diagnosis of chronic venous disease is based on anamnesis, clinical symptoms and diagnostic tests. Today, duplex ultrasound is the gold standard for the diagnosis of CVI. The most widely used classification system for the classification of CVI is the CEAP classification system, which includes clinical, etiological, anatomical and pathophysiological effects and stages. In this classification, CEAP stands for; C: Clinical appearance, E: Etiological factors, A: Anatomical distribution, P: Pathophysiological condition. In general, C (clinical features)-classification is used in daily clinical practice. Insufficiency of the muscle pump includes not only calf muscle insufficiency but also respiratory muscle insufficiency. The diaphragm is a dome-shaped musculofibrous layer that separates the thorax and abdomen. The diaphragm, which acts as the main inspiratory muscle, creates a suction effect on the inferior vena cava during inspiration and expiration, allowing more blood flow from the lower extremities to the heart. Changes in pressure in the thoraco-abdominal region directly affect venous flow. Inspiration increases negative intrathoracic pressure, causing blood to be sucked into the thorax. Simultaneously, the diaphragm contracts and the abdominal veins are compressed. These changes in intrathoracic and intraabdominal pressures that occur with respiration help venous return by preventing retrograde flow in the veins. It has been shown that the respiratory cycle affects venous return in healthy individuals, and that the flow rate in the femoral vein increases with deep inspiration. However, no study has been found examining the relationship between disease severity, edema, pain, respiratory muscle strength, respiratory functions, aerobic capacity, lower extremity strength and quality of life in individuals with chronic venous insufficiency. For this reason, since the relationship between disease severity, disease symptoms, respiratory functions, aerobic capacity and quality of life in individuals with chronic venous insufficiency is unknown, this study aimed to clarify it.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with chronic venous insufficiency
* Agreeing to participate in the study
* Being 18 years of age or older

Exclusion Criteria:

* Presence of arterial diseases
* Presence of advanced cardiorespiratory diseases
* Presence of acute ulcers (< 3 months) and diabetic ulcers
* Being pregnant
* Presence of deep vein thrombosis
* Presence of active infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with chronic venous insufficiency volunteered to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Disease severity | From July 2023 to May 2024
  The disease severity (CEAP scores) of the individuals referred to the study were determined by the cardiovascular surgeon.

SECONDARY OUTCOMES:
Evaluation of Lower Extremity Strength | From July 2023 to May 2024
  The 30-second Sit-to-Stand Test was used on a chair to determine lower extremity strength and functional mobility. Rikli et al. designed a 30-second sit-to-stand test in 1999 to evaluate individuals' dynamic balance and physical fitness lower extremity neuromuscular function levels. During the test, the individual sat on a chair without back support, arms crossed over the body, which was the initial sitting position. Then, the individual stood up and sat down repeatedly for 30 seconds. The total number of correct standing ups during this period was recorded. A higher number of repetitions indicates better physical performance. Performing less than 10 repetitions of the movement in 30 seconds indicates lower extremity weakness.
Assessment of aerobic capacity | From July 2023 to May 2024
  The 6-minute walking test was performed according to ATS criteria and twice on the same day, half an hour apart. Before the test, the subjects rested for at least 10 minutes, and before and after the test, oxygen saturation, heart rate, blood pressure, respiratory rate, dyspnea perception, fatigue and leg fatigue were recorded. Oxygen saturation was assessed using a portable pulse oximeter, heart rate using a heart rate monitor, blood pressure using a sphygmomanometer, respiratory rate using a count of the breaths taken per minute, and fatigue, leg fatigue and dyspnea perception using the Modified Borg Scale. The starting and ending points in the corridor where the test would be performed were determined and marked with cones. The subjects were asked to walk as fast as they could at their own walking speed for 6 minutes on a 30-meter straight corridor. In order to encourage the subjects, standard expressions were used for each minute during the test and the 6-MWT distance was recorded
Evaluation of respiratory functions | From July 2023 to May 2024
  A spirometer was used to evaluate respiratory functions. Before the test, individuals rested for 15 minutes and during the rest, participants were told how to do the test, how to use a mouthpiece, when to inhale and exhale, and how to complete the test with maximum effort, and then they were shown a practical demonstration. While individuals were sitting in a comfortable position in a chair with a back, a clip was placed on their noses and they were asked to bite the mouthpiece with their teeth and close their lips so that they would not allow air to escape. During the test, individuals were asked to exhale until there was no air left in their lungs and they were allowed to follow the time on the monitor. The tests were to be performed by the participants at least 3 times and it was ensured that the expiration time was at least 6 seconds and the plateau time was 1 second.
Respiratory muscle strength assessment | From July 2023 to May 2024
  Respiratory muscle strength was assessed with a spirometer. The pressure was recorded during a few seconds of maximal inspiration (Müller maneuver) or expiration (Valsalva maneuver) through the mouth. Maximum static inspiratory pressure was measured by having the patients take a rapid and deep inspiration at the residual volume after maximum expiration. Maximum static expiratory pressure was measured by having the patients take a rapid and deep expiration at the total lung capacity after maximum inspiration. The tests were performed in the sitting position using a nose clip. The patients were verbally encouraged to achieve the best strength. The measurement was repeated until a valid value was obtained in the patients. If there was a difference of more than 5% or 5 cmH₂O between the consecutive measured values, the measurement was repeated.
Quality of life assessment | From July 2023 to May 2024
  The Chronic Venous Insufficiency Quality of Life Questionnaire (CIVIQ) was used to assess quality of life. The questionnaire consists of 20 questions specific to Chronic Venous Insufficiency. It consists of 4 parameters questioning physical, psychological, social status and pain. Each question is scored according to a 5-item Likert scale. Higher scores indicate better quality of life. The Turkish validity and reliability study was conducted by Özdemir et al.
Pain Assessment | From July 2023 to May 2024
  Pain intensity was measured with the Numerical Rating Scale (SDS). The maximum level of pain felt at rest and during activity was scored from 0 to 10. A value of "0" indicates no pain, and a value of "10" indicates pain of the worst intensity. The reliability and validity of the SDS was proven by Cleland et al., and the intraclass correlation coefficient (ICC) value was reported as 0.76.
Edema Assessment | From July 2023 to May 2024
  The edema in the lower extremity was assessed by measuring the circumference with a tape measure. Each leg was recorded separately and the difference was calculated. A flexible, non-elastic, 7 mm wide standard tape measure with a sensitivity level of 0.1 cm was used in circumference measurements. The "0" (zero) end of the tape measure was wrapped around the area to be measured, with the other end in the left hand and the number on the "0" (zero) point noted. During the measurement, care was taken to ensure that the "0" (zero) point of the tape measure and the measurement number were side by side, not on top of each other, and the measurement was performed with the patient in the supine position in order to ensure standardization in each measurement. The circumference measurement values for each individual were converted to volumetric measurements by placing them in the Frustrum formula (truncated cone method).

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Çinar Özdemir, Prof.Dr, Principal Investigator — İzmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Karabağlar/İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Ozdemir OC, Tonga E, Tekindal A, Bakar Y. Cross-cultural adaptation, reliability and validity of the Turkish version of the Chronic Venous Disease Quality of Life Questionnaire (CIVIQ-20). Springerplus. 2016 Mar 31;5:381. doi: 10.1186/s40064-016-2039-2. eCollection 2016. PMID 27066388
- [Background] Kwon OY, Jung DY, Kim Y, Cho SH, Yi CH. Effects of ankle exercise combined with deep breathing on blood flow velocity in the femoral vein. Aust J Physiother. 2003;49(4):253-8. doi: 10.1016/s0004-9514(14)60141-0. PMID 14632624
- [Background] Osada T, Katsumura T, Hamaoka T, Murase N, Naka M, Shimomitsu T. Quantitative effects of respiration on venous return during single knee extension-flexion. Int J Sports Med. 2002 Apr;23(3):183-90. doi: 10.1055/s-2002-23177. PMID 11914981
- [Background] Tracz E, Zamojska E, Modrzejewski A, Zaborski D, Grzesiak W. Quality of life in patients with venous stasis ulcers and others with advanced venous insufficiency. Holist Nurs Pract. 2015 Mar-Apr;29(2):96-102. doi: 10.1097/HNP.0000000000000072. PMID 25658932